CLINICAL TRIAL: NCT05167097
Title: Updating Risk (DFG 441551024) - Work Package 2 - Mindsets Influence the Effectiveness of a Brief Intervention
Brief Title: Mindsets and the Effectiveness of a Brief Intervention - Replication
Acronym: MindsetBI-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Lucas Keller, Principal investigator, University of Konstanz
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: Mindset BI Replication 2021
Record Dates: First submitted 2021-10-29; First posted 2021-12-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Drinking; Cannabis Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking only applies to mindset manipulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Deliberative Mindset (Experimental): Participants receive a paper/pencil questionnaire that evokes a deliberative mindset. The questionnaire asks participants to deliberate upon the positive and negative short- and long-term consequences of acting vs. not acting toward a goal. This procedure is based on previous research on the mindset theory of action phases.
  Interventions: Other: Mindset Intervention
- Implemental Mindset (Experimental): Participants receive a paper/pencil questionnaire that evokes an implemental mindset. The questionnaire asks participants to plan the when, where, and how of taking five steps toward a goal. This procedure is based on previous research on the mindset theory of action phases.
  Interventions: Other: Mindset Intervention
- Decisional Balance BI (Experimental): Participants receive the ASSIST-linked Brief Intervention via an interview with a trained interventionist. The decisional balance element describes Steps 6-9 of the ten steps of the manual. They include probing for the positive and negative sides of alcohol consumption, weighing them against each other, focusing on the negative sides, and asking participants how concerned they are regarding the negative sides.
  Interventions: Other: ASSIST-linked Brief Intervention
- No Decisional Balance BI (Experimental): Participants receive the ASSIST-linked Brief Intervention via an interview with a trained interventionist. This is the short-form of the ASSIST-linked Brief Intervention. It drops the decisional balance element that is described above.
  Interventions: Other: ASSIST-linked Brief Intervention
- Control Group (Other): Participants perform a filler task in the control group, crossing out a specific letter in paragraphs of nonsense text.
  Interventions: Other: Mindset Intervention

INTERVENTIONS:
Other: ASSIST-linked Brief Intervention — WHO's ASSIST-linked Brief Intervention (with and without Steps 6-9, the decisional balance element)
  Arms: Decisional Balance BI; No Decisional Balance BI
Other: Mindset Intervention — Standard mindset manipulation as used in research by Peter M. Gollwitzer and colleagues
  Arms: Control Group; Deliberative Mindset; Implemental Mindset

SUMMARY:
Brief Interventions (BI) based on Motivational Interviewing are effective in reducing alcohol use. In this study, the investigators test the hypothesis that mindsets increase the positive effects of BI among a student sample of risky drinkers.

Subjects will be students with risky alcohol use as identified by the AUDIT. All participants receive the World Health Organization's (WHO) ASSIST-linked BI in one of two forms. Either with or without a decisional balance element (Steps 6-9 from the ten steps of the intervention). Before the ASSIST-linked BI, participants are randomly assigned to one of three mindset conditions. They either deliberate upon an unsolved problem (deliberative mindset), plan the implementation of a set goal (implemental mindset), or perform a control task (control condition).

The investigators measure the change in alcohol-related risk perceptions, treatment motivation, and alcohol drinking as assessed via the timeline follow-back method. The investigators also assess THC consumption during the study.

DETAILED DESCRIPTION:
In this study, the investigators will try to advance our understanding of the effects of mindset inductions for coping with motivational interventions in hazardously drinking students. In an earlier study, the investigators found an interactive effect of implemental mindsets with motivational interviewing on actual risk behavior but not risk perception. The investigators will target potential underlying processes (e.g., resistance to change, commitment), as well as compensation and generalization effects by including the assessment of consumption of alternative risky substances.

The investigators target consumption-related risks and address interactions between mindsets and motivational interviewing. Combining a mindset induction with a Screening and Brief Intervention tool in which the risk status of the individual was assessed, and the interventionist provided feedback, conducted a decisional balance exercise, and used techniques from motivational interviewing, the investigators found effects on risk taking but not risk perception. Neither general risk taking in the subscales of the Domain-Specific Risk-Taking Scale nor alcohol-related risk perception in a specific questionnaire was significantly affected by our manipulations. Still, participants in an implemental mindset managed to reduce their monthly alcohol consumption on average by about 7 to 8 standard units (equates to roughly five glasses of wine) while participants in a deliberative mindset actually increased their alcohol consumption by a similar amount. The investigators want to replicate the earlier findings while simultaneously enriching our research design with a) a control condition to test whether the implemental mindset decreased drinking, the deliberative mindset increased drinking, or both happened concurrently, b) test for compensation and/or generalization effects by including the assessment of another substance, namely Tetrahydrocannabinol (THC), to see if participants may compensate their reduced alcohol consumption by enhanced consumption of substitutes or if they can self-regulate the consumption of both, and c) to test whether the decisional balance element of the ASSIST-linked brief intervention is driving the differences between mindsets.

Design. The experiment follows a 3 between (Mindset: deliberative vs. implemental vs. control) x 2 between (Brief Intervention: short-form [without decisional balance] vs. long-form [with decisional balance]) factorial experimental design. Main dependent variables are the Timeline Followback (TLFB)-based self-reports of substance consumption, alcohol-related risk perception, and moderating/mediating variables related to the brief intervention itself (e.g., commitment, openness, resistance to change).

Hypotheses. In the control condition, the investigators expect to see similar results to earlier work on the effectiveness of motivational interviewing in reducing alcohol. In the deliberative and implemental mindset condition, however, the investigators expect to see a more nuanced picture, similar to our previous experiment. To better disentangle this, the investigators will include specific resistance and commitment ratings during the brief intervention session after the personalized feedback and after the decisional balance exercise that follows, the two subsequent parts of the brief intervention. The investigators hypothesize that deliberative mindset participants would show low resistance during personalized feedback but high resistance after the decisional balance exercise, and the opposite pattern for commitment. Implemental mindset participants, on the other hand, are expected to show the opposite pattern for resistance and commitment after the decisional balance exercise; it remains unclear, however, how this group will respond to the personalized feedback procedure. Furthermore, the investigators want to explore whether the reduction/increase in consumption is specific to the one substance that is addressed in the brief intervention or whether regulation of consumption also affects alternative substances in terms of generalization or compensation. The investigators use THC as a model substitute because of the high prevalence (e.g., 64% in an earlier study.

Procedure. The procedure will be very similar to our previous experiment. Participants will first be screened using an online questionnaire, and only at-risk drinking individuals (as indicated by the AUDIT) will be invited to the first lab session. Participants then receive the mindset manipulation. The investigators will ensure that the interventionist will be blind to the participants' mindset condition and that the mindset manipulation will involve a problem or project that is not related to substance use. Thereafter, the interventionist will assess the individuals' risk behavior regarding a set of substances (using the WHO's ASSIST manual) in an interview setting and will give the participants individualized feedback on their consumption (i.e., the first phase of the brief intervention). The interventionist will then conduct a motivational interview about the participants' personal alcohol consumption (i.e., the second phase of the brief intervention). Afterward, the interventionist will rate how resistant the participants behaved during the intervention. Thereafter participants report their alcohol and THC consumption for the last four weeks using the TLFB and fill out a series of questionnaires. Four weeks later, participants are back for a second lab session in which they again fill out the same battery of questionnaires to assess their (alcohol-specific) risk perception and to assess their alcohol and THC consumption, again using the TLFB.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT > 8 in a prescreening

Exclusion Criteria:

* Alcohol use disorder or substance use disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Use | 4 weeks before and 4 weeks after the intervention
  Assessed via the Timeline Followback method
Change in THC Use | 4 weeks before and 4 weeks after the intervention
  Assessed via the Timeline Followback method

SECONDARY OUTCOMES:
Change in Individual Risk Perception (general) | In between two sessions (i.e., 4 weeks)
  Assessed via a single question asking participants how willing they are to take risks (on a 11-point scale)
Change in Individual Risk Perception (alcohol-specific) | In between two sessions (i.e., 4 weeks)
  Assessed via the Questionnaire to assess alcohol-related risk perception

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Keller, PhD, Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
In an anonymized data file on a public repository.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon submission to a peer-reviewed journal and for at least 7 years as advised by the American Psychological Association
Access Criteria: Anonymized data will be accessible to anyone with a link to the data file in the publication.